CLINICAL TRIAL: NCT02138734
Title: A Study of Intravesical Bacillus Calmette-Guerin (BCG) in Combination With ALT-803 (N-803) in Patients With Non-Muscle Invasive Bladder Cancer
Brief Title: A Study of Intravesical BCG in Combination With ALT-803 in Patients With Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-01-14; QUILT-2.005
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: antitumor; BCG; bladder cancer; cancer; immunotherapy; instillation; interleukin-15; intravesical; naive; non-muscle invasive; transitional cell carcinoma; ALT-803; N-803
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Single arm phase Ib.
  Two-arm phase IIb, two-cohort: each randomized 1:1 via randomization scheme stratified by disease and ECOG status.
  Cohort A: patients with CIS disease (with or without Ta/T1); planned enrollment = 366 Cohort B: patients with high-grade papillary disease (Ta/T1 only); planned enrollment = 230
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-803+BCG (Experimental): (Phase Ib and IIb) for BCG-naive patients
  Interventions: Biological: BCG+N-803( 50mg BCG/ Instillation+ N-803( 400 μg/instillation). )
- BCG alone (Active Comparator): (Phase IIb) for BCG-naive patients
  Interventions: Biological: BCG( 50mg/Instillation)

INTERVENTIONS:
Biological: BCG+N-803( 50mg BCG/ Instillation+ N-803( 400 μg/instillation). ) — BCG and N-803 will be mixed together (with saline) and administered via intravesical instillation weekly for 6 consecutive weeks for induction. Phase IIb includes maintenance treatment consisting of BCG+N-803 for 3 consecutive weeks at 3, 6, 12, 18, 24,30 and 36 months.
  An additional 6 week re-induction of BCG+N-803 for patients with eligible disease at 3 months in phase IIb is included.
  Arms: N-803+BCG
Biological: BCG( 50mg/Instillation) — BCG will be administered via intravesical instillation weekly for 6 consecutive weeks for induction. Phase IIb includes maintenance treatment consisting of BCG for 3 consecutive weeks at 3, 6, 12, 18, 24, 30 and 36 months.
  An additional 6 week re-induction of BCG for patients with eligible disease at 3 months in phase IIb is included.
  Arms: BCG alone

SUMMARY:
This is a Phase Ib/IIb, randomized, two-cohort, open-label, multicenter study of intravesical N-803 plus BCG versus BCG alone, in BCG naïve patients with high-grade NMIBC.

DETAILED DESCRIPTION:
The study includes a dose escalation phase (phase Ib) and an expansion phase (phase IIb).

In the phase Ib, patients will be treated with intravesical N-803 in combination with BCG. The purpose of the phase Ib portion of the study is to evaluate the safety, identify the Maximum Tolerated Dose (MTD) of N-803 and determine the Recommended Dose (RD) level of N-803 in combination with BCG for the phase IIb expansion.

In the phase IIb expansion, patients will be randomized to receive either intravesical N-803 in combination with BCG or BCG alone. Patients will be enrolled into one of two study cohorts (Cohort A and Cohort B). These will be two independent study cohorts, evaluated separately for treatment efficacy.

ELIGIBILITY:
Inclusion Criteria

1. Histologic confirmation of non-muscle invasive bladder cancer of the transitional cell carcinoma high-grade subtype (mixed histology tumors allowed if transitional cell histology is predominant histology).

   1. Cohort A: Histologically confirmed CIS (with or without Ta/T1 disease); Cohort B: Histologically confirmed high-grade papillary disease (Ta/T1 only).
   2. Patients are eligible if the diagnostic biopsy was done within 3 months of treatment start and a cystoscopy demonstrating no resectable disease was done within 6 calendar weeks (inclusive of 48 days) of treatment start (residual CIS is acceptable; patients with T1 disease must undergo repeat resection if muscularis propria is not present in each biopsy sample). Patients with high-grade Ta and/or T1 disease should have complete resection before study treatment.
   3. Upper tract imaging within 6 months prior to study entry must not be suspicious for upper tract malignancy.
2. Currently eligible for intravesical BCG therapy.
3. Age ≥ 18 years.
4. Performance status: ECOG performance status of 0, 1, or 2.
5. BCG-naive disease as defined as either of the following:

   1. Have not received prior intravesical BCG; or
   2. Previously received BCG, but stopped receiving more than 3 years before date of randomization.
6. Laboratory tests performed within 21 days of treatment start:

   1. Absolute lymphocyte count ≥ Institutional lower limit of normal
   2. Absolute neutrophil count (AGC/ANC) ≥ 1,000/μL
   3. Platelets ≥ 100,000/µL [Patients may be transfused to meet this requirement]
   4. Hemoglobin ≥ 8 g/dL [Patients may be transfused to meet this requirement]
   5. Calculated glomerular filtration rate (GFR*) >40 mL/min or Serum creatinine ≤ 1.5 x ULN
   6. Total bilirubin ≤ 2.0 X ULN
   7. AST, ALT, ALP ≤ 3.0 X ULN
7. Adequate pulmonary function without any clinical sign of severe pulmonary dysfunction. PFT > 50% FEV1 if clinically indicated by the investigator.
8. Negative serum pregnancy test if female and of childbearing potential (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized).
9. Female participants of childbearing potential must adhere to using a medically accepted method of birth control prior to screening and agree to continue its use during the study or be surgically sterilized (e.g., hysterectomy or tubal ligation) and males must agree to use barrier methods of birth control while on study.
10. Provide signed informed consent and HIPPA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations.

    * using the following Cockcroft-Gault equation to calculate the eGFR for this study: eGFR in mL/min = {(140-age in years) x (weight in kg) x F}/(serum creatinine in mg/dL x 72) Where F =1 if male; and 0.85 if female

Exclusion Criteria

1. Prior BCG treatment or known hypersensitivity to BCG. Patients who have received more than a single-dose post-operative treatment of mitomycin-C or gemcitabine following the most recent screening TURBT/biopsy are excluded.
2. Concurrent use of other investigational agents (not including FDA-authorized drugs for the prevention and treatment of COVID-19).
3. History of or evidence of muscle-invasive, locally advanced, metastatic and/or extravesical bladder cancer or any other cancer within the past 5 years, except: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage 1 or 2 cancer from which the patient is currently in complete remission, or stable prostate cancer (under active surveillance or hormone control).
4. Symptomatic congestive heart failure (CHF), NYHA (New York Heart Association) Class III or IV or other clinical signs of severe cardiac dysfunction.
5. Severe/unstable angina pectoris, or myocardial infarction within 6 months prior to study entry.
6. History or evidence of uncontrollable CNS disease.
7. Known HIV-positive.
8. Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
9. Concurrent febrile illness, active urinary tract infection, active tuberculosis, a history of hypotension or anaphylactic reactions.
10. Ongoing chronic systemic steroid therapy required (>10 mg oral prednisone daily or equivalent).
11. Women who are pregnant or nursing. Female patients of childbearing potential must have a negative pregnancy test and must adhere to using a medically acceptable method of birth control prior to screening and agree to continue its use during the study and for 30 days after the last dose of study drug, or be surgically sterilized (e.g., hysterectomy or tubal ligation). Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Males must agree to use barrier methods of birth control while on study and for 90 days post last dose of study drug.
12. Psychiatric illness/social situations that would limit compliance with study requirements.
13. Other illness that in the opinion of the investigator would exclude the patient from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2014-07-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | 6 Months
  Patients in Cohort A: compare complete response rate between treatment arms using cystoscopy, confirmatory bladder biopsy and urine cytology.
Disease Free Survival (DFS) | 13 Years and 3 Months
  Patients in Cohort B: compare disease-free survival between treatment arms using
  cystoscopy, confirmatory bladder biopsy and urine cytology.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 13 Years and 3 Months
  For phase IIb, Cohorts A & B: Time from randomization to disease progression or death.
Overall survival | 13 Years and 3 months
  Time from randomization to death resulting from any cause to determine survival.
Disease specific survival | 13 Years and 3 months
  For phase IIb, Cohorts A & B: Time from randomization to death resulting from bladder cancer.
Time to disease worsening | 13 Years and 3 Months
  For phase IIb, Cohorts A & B: Cystectomy or change in therapy indicative of more advanced disease, including systemic chemotherapy or radiation therapy.
Cystectomy Free Rate | 13 years and 3 months
  Cystectomy-free rate will be calculated for each treatment group as the ratio of the number of subjects who don't have documented cystectomy in the database divided by the number of subjects in the ITT (Intent to treat) population.
Safety Profile: Number and severity of treatment emergent AEs [Time Frame: 39 Months] | 39 Months
  For phase Ib and phase IIb: Number of participants with TEAEs as assessed by CTCAE v4.03.
Duration of Complete Response | 13 Years and 3 months
  To assess the duration of CR of patients treated with N-803 plus BCG compared to patients treated with BCG alone.
Complete Response Rate( All Recurrent Bladder Cancer Including Low Grade Ta Disease) | 13 Years and 3 months
  To assess the CR rate (all recurrent bladder cancer including low grade Ta disease) of patients treated with N-803 plus BCG compared to patients treated with BCG alone.
Long Term Complete Response Rate | 13 years and 3 Months
  To assess the long-term CR rate (as determined by the Investigator) following completion of QUILT-2.005 phase 2b.
Duration of Complete Response ( All Recurrent Bladder Cancer Including Low Grade Ta Disease) | 13 Years and 3 months
  Time from the date of first CR (All Recurrent bladder cancer including low grade Ta Disease) to the date of evidence that the subject no longer meets the definition for CR.
Cohort B: Disease Free Survival Rate | 36 Months
  To assess DFS rate at 12, 18, 24, 30, and 36 months. The time from randomization until recurrence of high-grade Ta (excluding low grade Ta) or any grade T1, CIS, disease progression, cystectomy, change in therapy indicative of more advance disease or death (any cause), whichever occurs first.
Cohort B: Disease Free Survival | 13 Years and 3 Months
  DFS was assessed in the following groups:
  1) All recurrent bladder cancer, including low grade Ta disease the time from randomization until recurrence of any grade Ta (including low grade Ta) or any grade T1, CIS, disease progression, cystectomy, change in therapy indicative of more advanced disease, or death (any cause), whichever occurs first 2) Patients who have high-grade Ta, low-grade T1, or CIS at 3-months and received re-induction, and have no evidence of > low-grade Ta disease at 6-months will be considered disease-free from randomization until a second recurrence > low-grade Ta 3) Patients who have high-grade Ta, low-grade T1, or CIS at 3-months and received re-induction, and have no evidence of any disease (including low grade Ta) at 6-months will be considered disease-free from randomization until a second recurrence ≥ low grade Ta.
Vital signs and clinical laboratory assessment | 36 Months
  Vital signs include heart rate, systolic and diastolic blood pressures, respiration rate, and body temperature. Labs include the following: complete blood count with differential, complete metabolic panel, and urinalysis.
Long Term Follow Up(LTFU) data from subjects who were treated | 10 Years after treatment period visits
  Yearly collection of LTFU data, which includes the following: survival status, bladder cancer status (high or low grade), cystoscopy results including number of cystoscopies done for each subject, biopsy results, upper tract evaluations, posttherapies and responses and outcomes of posttherapies, urine cytology results, and other medical history or treatments, if available, related to bladder cancer.

OTHER OUTCOMES:
Exploratory Endpoints- Immunogenicity: Serum level of anti-N-803 in patient samples | 36 Months
  For phase Ib and IIb Measures the serum level of anti-N-803 in patient samples.
Quality of Life Endpoint | 39 Months
  Quality of Life (QoL) as assessed by the European Organization for Research and Treatment of Cancer (EORTC) questionnaires for patients with cancer (QLQ-C30) and for patients with NMIBC (QLQ-NMIBC24).
Exploratory Endpoints- Whole Slide Images (Baseline and any on-study biopsy) | 39 Months
  For Phase IIb

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Reddy, MD, Study Director — ImmunityBio, Inc.
Locations (80):
- United States (53):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Arkansas Urology, Little Rock, Arkansas
  - Hoag Cancer Center, Irvine, California
  - UCLA Department of Urology, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - Skyline Sherman Oaks, Sherman Oaks, California
  - Skyline Urology, Torrance, California
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Memorial Healthcare System, Hollywood, Florida
  - Advanced Urology Institute, Oxford, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Florida Urology Partners, Riverview, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Associated Urological Specialists, Chicago, Illinois
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - UroPartners, Glenview, Illinois
  - Urology of Indiana, Carmel, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Urology, Royal Oak, Michigan
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Urology Group of New Mexico (AccumetRx Clinical Research), Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - Integrated Medical Professionals, New York, New York
  - NYU Langone Health, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Lowcountry Urology Clinics, North Charleston, South Carolina
  - Erlanger Health, Chattanooga, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Urology Partners of North Texas, Arlington, Texas
  - Texas Oncology, Austin, Texas
  - Urology Austin, PLLC, Research Department, Austin, Texas
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Potomac Urology, Alexandria, Virginia
  - Virginia Urology, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - University of Washington School of Medicine, Seattle, Washington
- India (26):
  - HCG Cancer Centre, Visakhapatnam, Andhra Pradesh
  - Darakh Nursing Home and Kidney Stone Centre, Aurangabad, Maharashtra
  - Kidney Centre Jasleen Hospital, Nagpur, Maharashtra
  - Indriyani Hospital & Cancer Institute, Pune, Maharashtra
  - HCG Manavata Cancer Centre, Mumbai, Nashik
  - Erode Cancer Centre, Erode, Tamilnadu. India
  - Pi Health Cancer Hospital, Hyderabad, Telangana
  - Swami Harshankaranand JI Hospital and Research Centre, Sunderpur, Varanasi
  - B J Medical College & Civil Hospital, Asarwa, Ahmedaba, Ahmedabad
  - Basavatarakam Indo American Cancer Hospital & Research Institute, Banjara Hills
  - HCG Bangalore, Bengaluru
  - SP Medical College and Hospital, Bikaner
  - Guru Govnid Singh Medical College and Hospital, Farīdkot
  - Muljibhai Patel Urological Hospital, Gujrāt
  - Binayak Multispecialty Hospital, Kolkata
  - Chittaranjan National Cancer Institute, Kolkata
  - KR Hospital, Mysuru
  - KMC Manipal, Nagar
  - Jasleen Hospital, Nagpur
  - Onco Life Cancer Center, Pune
  - Inamdar Hospital Pune, Pune
  - Urocare Hospital, Rajkot
  - All India Institute of Medical Sciences, Raipur, Rajpura
  - Uttar Pradesh University of Medical Sciences, Uttar
  - HCG cancer Centre, Vizag, Visakhapatnam
  - Apollo Vizag, Visakhapatnam
- SunningHill Hospital, Sandton, South Africa

REFERENCES:
- [Derived] Chamie K, Chang SS, Rosser CJ, Kramolowski E, Gonzalgo ML, Sexton WJ, Spilman P, Sender L, Reddy S, Soon-Shiong P. N-803 Plus BCG Treatment for BCG-Naive or -Unresponsive Non-Muscle Invasive Bladder Cancer: A Plain Language Review. Future Oncol. 2024;20(31):2307-2317. doi: 10.1080/14796694.2024.2363744. Epub 2024 Jul 2. PMID 38953850